CLINICAL TRIAL: NCT07295821
Title: Phase II, Single-arm Multicenter Study of Osimertinib Induction Before Radiotherapy and Maintenance in Chemo-ineligible or Refusing Patients With Stage III, Unresectable NSCLC and EGFR Mutation-positive Tumors
Brief Title: Osimertinib Induction and Maintenance for Chemo-ineligible Stage III Unresectable EGFR+ NSCLC: Single-arm Study
Acronym: NSCLC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D5167L00001
Record Dates: First submitted 2025-11-24; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Lung Cancer
Keywords: NSCLC
MeSH Terms: conditions — Lung Neoplasms | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Osimertinib as Induction Therapy Prior to Radiotherapy and Maintenance (Experimental): 80 mg Osimertinib QD
  Interventions: Drug: Osimertinib

INTERVENTIONS:
Drug: Osimertinib — 80 mg Osimertinib QD

SUMMARY:
The purpose of this study is to measure efficacy and safety of osimertinib as induction therapy prior to curative intent RT and maintenance osimertinib in chemotherapy ineligible or refusal adult patients with Stage III, unresectable NSCLC with common EGFR mutations (exon 19 deletion or L858R).

DETAILED DESCRIPTION:
Study details include:

* The study duration will be approximately 13 months for recruitment and 2 years of follow up from the last patient's initiation into the study.
* The induction treatment with osimertinib will be up to12 weeks, followed by 6 weeks of RT treatment and osimertinib maintenance treatment until disease progression or death.
* The visit frequency will be once after 12 weeks during the induction treatment period, every 3 weeks during the RT period (daily visits for RT), and every 12 weeks during the osimertinib maintenance treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be ≥ 18 years or the legal age of consent in the jurisdiction in which the study is taking place, at the time of signing the informed consent form.
2. Participants with histologically documented NSCLC of predominantly nonsquamous, squamous, and adenosquamous pathology who present with locally advanced, unresectable (Stage III, according to Version 8 of the IASLC Staging Manual in Thoracic Oncology) disease. It is recommended but not required that except for overt cT4 disease, nodal status N2, or N3 should have been proven by biopsy, via endobronchial ultrasound, mediastinoscopy, thoracoscopy, or in absence of biopsy, should have been confirmed with whole body contrast-enhanced CT.
3. Participants who had recurred from Stage I/II/III after complete surgery or had gross incomplete resections can be included if they didn't receive treatment with any chemotherapy, radiation therapy, immunotherapy, targeted therapy, or investigational agents.
4. Participants with availability of the EGFRm test results confirming that the tumor harbors 1 of the 2 common EGFR mutations known to be associated with EGFR-TKI sensitivity (Ex19del, L858R), either alone or in combination with other EGFR mutations including de novo T790M
5. WHO performance status of 0, 1 or 2 with no deterioration over the previous 2 weeks prior to baseline at screening and prior to first dose.
6. Participants who are eligible for and planning to undergo RT treatment per physician assessment.
7. Participant refusal or ineligible for chemotherapy per physician assessment.
8. Minimum life expectancy of > 12 weeks at Day 1.
9. At least one lesion that can be accurately measured at baseline as ≥ 10 mm in the longest diameter (except lymph nodes, which must have short axis ≥ 15 mm) with CT or MRI and is suitable for accurate repeated measurements.
10. Capable of giving signed informed consent as described which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.

Exclusion Criteria

1. Any presence of small cell and mixed small-cell and non-small cell histology.
2. Past medical history of ILD, drug-induced ILD, radiation pneumonitis that required steroid treatment, or any evidence of clinically active ILD.
3. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, which in the investigator's opinion makes it undesirable for the participant to participate in the trial or which would jeopardize compliance with the protocol, or active infection.
4. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of osimertinib.
5. History of another primary malignancy except for malignancy treated with curative intent with no known active disease ≥ 2 years before the first dose of study intervention and of low potential risk for recurrence. Exceptions include adequately resected non-melanoma skin cancer and curatively treated in situ disease. Patients who have received RT with overlapping fields (eg, cured breast cancer) should be excluded.
6. Patient meets any of the following cardiac criteria: Mean resting QTc > 470 msec, obtained from 3 ECGs, using the screening clinic ECG machine-derived QTc value.
7. Inadequate bone marrow reserve or organ function.
8. Any unresolved toxicities from prior therapy greater than CTCAE Grade 1 at the time of starting study treatment with the exception of alopecia and Grade 2 prior platinum-therapy related neuropathy. Prior treatment with any chemotherapy, radiation therapy, immunotherapy, targeted therapy, or investigational agents for locally advanced, unresectable Stage III NSCLC. Prior surgical resection (ie, Stage I, II, or III) with no systemic treatment with residual disease or a recurrence is permitted.

11 Prior exposure to EGFR-TKI therapy. 12 Major surgical procedure (excluding placement of vascular access) or significant traumatic injury within 4 weeks of the first dose of study intervention or an anticipated need for major surgery during the study.

13 Participation in another clinical study with a study intervention or investigational medicinal device administered in the last 4 weeks.

14 History of hypersensitivity to active or inactive excipients of osimertinib or drugs with a similar chemical structure or class to osimertinib.

15 History of hypersensitivity to active or inactive excipients of RT. 16 Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).

17 Judgment by the investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions, and requirements.

18 Previous enrolment in the present study. Rescreening of individuals who were screen failures is allowed.

19 For females only - currently pregnant (confirmed with positive pregnancy test) or breastfeeding.

20 Patients should refrain from breastfeeding from enrolment throughout the study and until 6 weeks after last dose of study intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-03-09 (Estimated); Primary Completion 2029-05-30 (Estimated); Study Completion 2029-05-30 (Estimated)

PRIMARY OUTCOMES:
PFS (Progression-Free Survival) | Assessed from date of first dose to progression (up to a maximum of approximately 2 years)
  PFS is defined as the time from date of first dose until progression per RECIST 1.1 as assessed by the investigator at the local site, or death due to any cause.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | Assessed during the induction phase of the study, scans are carried out at week 12 (plus or minus visit window).
  DCR is defined as the percentage of subjects who have a best overall response of CR or PR or SD (at 12 weeks) as determined by the investigator at the local site per RECIST 1.1.
Overall Survival (OS) | Assessed from first dose to end of study or death (up to a maximum of approximately 2 years)
  OS is defined as time from date of first dose until the date of death due to any cause.

OTHER OUTCOMES:
AEs | From signing ICF to 28 days after last dose or end of study (up to a maximum of approximately 2 years)
  To assess the safety of osimertinib used as an induction therapy prior to RT and maintenance osimertinib treatment by assessment of AEs in patients with unresectable EGFRm NSCLC

CONTACTS AND LOCATIONS:
Locations (17):
- China (17):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Foshan
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Harbin
  - Research Site, Hefei
  - Research Site, Jinan
  - Research Site, Kunming
  - Research Site, Nanchang
  - Research Site, Qingdao
  - Research Site, Shanghai
  - Research Site, Taiyuan
  - Research Site, Wenzhou
  - Research Site, Xuzhou

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trails via the request portal.
  All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrails.pharmacm.com/ST/Submission/Disclosure.
  Indicates that AZ accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrails.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in approved sponsored tool. Signed Data Sharing Agreement(non-negotiable contract for data accessors)must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MES to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrails.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home